CLINICAL TRIAL: NCT05943483
Title: To Establish the Traditional Chinese Medicine Based Intelligent Personal Health Care System
Status: Completed | Type: Observational
Sponsor: Sheng-Teng Huang (Other)
Responsible Party: Sponsor-Investigator, Sheng-Teng Huang, Attending physician, China Medical University Hospital
Organization: China Medical University Hospital (Other)
Other Study IDs: CMUH109-REC1-026
Record Dates: First submitted 2023-07-03; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Traditional Chinese Medicine Body Constitution

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All subjects: Subjects who filled out our modified CCMQ questionnaire
  Interventions: Other: CCMQ questionnaire

INTERVENTIONS:
Other: CCMQ questionnaire — Test subjects were required to fill out our modified CCMQ (Constitution in Chinese Medicine Questionnaire) Questionnaire.

SUMMARY:
Development of a New Generation Chinese Medicine Constitution Assessment Scale

DETAILED DESCRIPTION:
Development of a New Generation Chinese Medicine Constitution Assessment Scale:

A. Analyzing the existing CCMQ and BCQ questionnaire syntax. B. Redesigning the scale's question statements. C. Reintegrating the scale items and constitutional characteristics. D. Testing and evaluating the reliability and validity of the questionnaire, cross-assessing with diagnoses from experienced Chinese medicine practitioners.

E. Collecting feedback and reviewing modifications based on the responses from the general population questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 and under 85.
* Participants agreed to join the trial by fully understanding the purpose of the study and the entire trial process and then signed an informed consent.
* Able to fill out online questionnaire with any electronic device in person or under assistance

Exclusion Criteria:

* Age of subjects was under 18 or more than 85 years old.
* Participants who do not meet the above criteria
* Subjects were not willing sign the informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The enrolled normal subjects were confirmed by the Association and the research Principal Investigator (PI). Subjects between the ages of 18 and 85 were included. We collected all of the subjects' basic information and administered the Chinese Medicine Constitution Assessment Scale.
Sampling Method: Non-Probability Sample
Enrollment: 1918 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Constitution in Chinese Medicine Questionnaire(CCMQ)_modified version | On the 1 day of receipt
  Based on the analysis, we have identified nine different types of Traditional Chinese Medicine constitutions.

SECONDARY OUTCOMES:
Base Data Questionnaire | On the 1 day of receipt
  Included collection of basic data (age, BMI, gender, place of residence, education level, smoking status, alcohol drinking, betel nut chewing, exercise frequency, work shift jobs and bedtime), disease status.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, North District, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD are not planned to be shared